CLINICAL TRIAL: NCT06036641
Title: The Effects of Prolonged Head-Down Tilt Lithotomy Position on Lower Limb Haemodynamics in Adults Undergoing Minimally Invasive Abdominopelvic Surgery: An Intraoperative Observational Study
Brief Title: The Effects of Prolonged Head-Down Tilt Lithotomy Position on Lower Limb Haemodynamics
Acronym: HELP
Status: Recruiting | Type: Observational
Sponsor: University of Portsmouth (Other)
Collaborators: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Principal Investigator, Maria Perissiou, Senior Lecturer, University of Portsmouth
Other Study IDs: IRAS [287464]; CPMS ID - 56254 (Other: NIHR Clinical Research Network (NIHR CRN))
Record Dates: First submitted 2023-09-03; First posted 2023-09-14 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Compartment Syndrome Nontraumatic Lower Extremity
Keywords: Head Down Tilt Lithotomy; Minimally Invasive Surgery; Ischaemia Reperfusion Syndrome; Pathophysiology; Near Infrared Spectroscopy, NIRS; Robotic Assisted Laparoscopic Surgery; Well leg Compartment Syndrome
MeSH Terms: interventions — Laser-Doppler Flowmetry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Colorectal surgery: Individuals scheduled for colorectal surgery in the HDTL position
  Interventions: Device: NIRS monitoring; Device: Laser Doppler flowmetry; Other: Inflammatory and Oxidative stress biomarkers

INTERVENTIONS:
Device: NIRS monitoring — All participants will undergo NIRS monitoring of muscle and cerebral tissue oxygenation intraoperatively.
Device: Laser Doppler flowmetry — Cutaneous blood flow will be assessed intraoperatively via Laser Doppler flowmetry in all participants
Other: Inflammatory and Oxidative stress biomarkers — Blood samples will be taken to measure biomarkers of inflammation and oxidative stress at specific time points

SUMMARY:
During certain bowel surgeries for cancer (colorectal surgery), individuals frequently have to be placed in a head-down position to enable surgeons have optimal access to the cancer site. This position usually also involves bending the hips and knees while supporting the legs in stirrups. However, lying in this position for long periods of time can lower the flow of blood to the legs, which can potentially cause injury. This rare but severe consequence is called Well-Leg Compartment Syndrome (WLCS). If WLCS is not diagnosed quickly, it can lead to other difficult complications and a significant delay in recovery. Unfortunately, because the individual is under anaesthesia, diagnosis is delayed in many cases. There is very little information in the medical literature about how this damage to the legs progresses over the course of the surgery. To better understand how WLCS, how well blood vessels work during surgery will be assessed. The flow of blood and oxygen in the calf muscle will be assessed in 25 individuals placed in a head-down position during colorectal surgery. Likewise, blood samples will be obtained in order to measure the biological markers that may contribute to the development of WLCS.

DETAILED DESCRIPTION:
The development of lower limb compartment syndrome in the absence of trauma (known as well-leg compartment syndrome, WLCS) is a severe complication reported during prolonged pelvic surgery. WLCS is characterised by muscular ischaemia and secondary necrosis from the increase in hydrostatic pressure in a closed fascial compartment.

The aetiology of WLCS appears to be primarily related to ischaemia of the lower limbs after a prolonged period in the head-down tilt lithotomy (HDTL) position, which is commonly used to access the pelvis and perineum during urological, colorectal, and gynaecological surgery. Elevation of the lower limbs above the heart results in a ~2 mmHg drop in mean arterial pressure at the mid-calf for every 2.5 cm that the limbs are raised. These hemodynamic changes are accompanied by an increase in compartment pressures associated with limb elevation and are further exacerbated by a steep (>15°) head-down tilt. The outcome of these changes ultimately leads to the development of significant and (often unrecognised) intraoperative ischemia in the lower limbs.

Prolonged reductions in lower limb perfusion during HDTL can cause the development of localised tissue oedema, leading to marked intracompartmental hypertension, which is further exacerbated once the limbs are lowered and reperfusion of ischemic muscle occurs. This is a consequence known as ischaemic-reperfusion injury (IRI), a phenomenon where reperfusion per se may result in a local and systemic inflammatory response that may augment tissue injury in excess of that produced by ischaemia alone.

Microvascular injury is considered one of the major determinants of IRI, particularly due to increased permeability of capillaries and arterioles that lead to an increase in diffusion and fluid filtration across the tissues. Subsequently, activated endothelial cells produce more reactive oxygen species and less nitric oxide, and this imbalance results in a corresponding inflammatory response and increased oxidative stress, which if sufficiently severe lead to further lower limb muscle and nerve injury.

The incidence of WLCS is unpredictable and as the individual is anaesthetised, the diagnosis is delayed in many cases, so the residual motor-sensory deficit may be severe, even after fasciotomy. Although there are many published case reports of this condition, it is likely that many cases of WLCS go unreported, and some may be mild and escape clinical detection. However, in cases that have been reported, the incidence of permanent disability after the development of WLCS ranges from ≈30% to ≈100%.

The paucity of detailed observational studies into the effects of HDTL on lower limb haemodynamics and tissue oxygenation has restricted the ability of the clinical and scientific society to construct clinical strategies to minimise this complication. Identifying individuals with risk factors and increasing surveillance during surgery in these people may allow for early detection and decrease the morbidity and potential mortality associated with intraoperative WLCS.

The study aims to assess lower limb haemodynamics by measuring cutaneous blood flow, muscle and brain tissue oxygenation, inflammatory and oxidative stress biomarkers during pelvic surgery in patients placed in HDTL. This study has the potential to provide a better understanding of the pathogenesis of WLCS and add novel knowledge regarding its early diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Adults scheduled to undergo colorectal surgery in the HDTL position

Exclusion Criteria:

* History of myocardial infarction or cerebro-vascular events in the last 12 months
* Previous revascularisation procedure in their lower limbs
* BMI > 40 kg/m2
* Inability to give informed consent
* Other serious medical conditions, which in the opinion of study investigators, would interfere with safety or data interpretation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult individuals(18 years and above) scheduled to undergo surgery in the HDTL position at the Department of Colorectal Surgery, Queen Alexandra Hospital, Portsmouth Hospitals University NHS Trust.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cutaneous blood flow | baseline, during the surgery
  Change over time in cutaneous blood flow in the legs relative to a vascular occlusion test (VOT) during surgery in the HDTL position.

SECONDARY OUTCOMES:
Muscle tissue oxygenation | baseline, during the surgery
  Change over time in muscle tissue oxygenation in the lower limb relative to a vascular occlusion test (VOT) during surgery in the HDTL position.
Plasma interleukin-6 (IL-6) concentration | baseline, during the surgery
  Change over time in [IL-6] during surgery in the HDTL position.
Plasma Tumour Necrosis Factor Alpha (TNF-α) concentration | baseline, during the surgery
  Change over time in [TNF-α] during surgery in the HDTL position.
Plasma Superoxide Dismutase (SOD) concentration | baseline, during the surgery
  Change over time in [SOD] during surgery in the HDTL position.
Plasma Protein Carbonyl concentration | baseline, during the surgery
  Change over time in [protein carbonyl] during surgery in the HDTL position.
Plasma nitrate concentration | baseline, during the surgery
  Change over time in [nitrate] during surgery in the HDTL position.
Plasma nitrite concentration | baseline, during the surgery
  Change over time in [nitrite] during surgery in the HDTL position.
Mean arterial pressure (MAP) | baseline, during the surgery
  Change over time in MAP during surgery in the HDTL position.
Skin temperature | baseline, during the surgery
  Change over time in skin temperature during surgery in the HDTL position.
Brain tissue oxygenation | continuous measurement during the surgery
  Change over time in brain tissue oxygenation during surgery in the HDTL position.

CONTACTS AND LOCATIONS:
Overall Officials: Chukwuemeka C Uzoma, MBBS, Principal Investigator — University of Portsmouth; Maria C Perissiou, PhD, Principal Investigator — University of Portsmouth
Locations (1):
- Queen Alexandra Hospital, Portsmouth Hospitals University NHS Trust, Portsmouth, West Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: No